CLINICAL TRIAL: NCT06794723
Title: A Single-center, Randomized, Double-blind, Parallel-group, Placebo-controlled Trial of a Probiotic-based Intervention to Improve Glycemic Control in Pregnancies Complicated by Gestational Diabetes.
Brief Title: A Probiotic Based Intervention in Pregnancies Complicated by GDM
Acronym: ProbioGDM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Graeme Smith, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6043857
Record Dates: First submitted 2024-12-20; First posted 2025-01-27 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-01

CONDITIONS: Gestational Diabetes Mellitus (GDM); Microbiome, Human
Keywords: Microbiome; Gestational Diabetes; Probiotic; Glucose Control; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to probiotic intervention or placebo. The randomization will be stratified by gestational age at randomization (1) Early - 25+0 to 27+6 weeks and (2) Late - 28+0 to 31+6 weeks. Randomization will be done with random block sizes of 3 and 6.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the treatment arms, the study staff, the study participants, and the care provider will be blinded to study arm assignment and will remain blinded until 6 weeks postpartum. At the end of the 6-week visit, once all data collection for that visit is complete, participants and study staff will be unblinded to the group assignment. Participants will then be provided with the option of enrolling in the extension of the intervention until 6 months postpartum. If they consent, additional open label investigational product will be dispensed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): The investigational product is a 5-strain probiotic plus prebiotic natural health product.
  Interventions: Dietary Supplement: 5-strain probiotic plus prebiotic natural health product
- Placebo (Placebo Comparator): Identically appearing placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 5-strain probiotic plus prebiotic natural health product — The investigational product is a 5-strain probiotic plus prebiotic natural health product for patients with Type 2 diabetes. Other ingredients include oligofructose, grape food color, magnesium stearate, silica and a delayed release capsule.
  Recommended storage is in a refrigerated environment at approximately 4°C. The product should not be frozen. It is recommended that the product be used within 2 months after opening the bottle. Participants are asked to take 2 capsules daily with food, 1 in the morning and 1 in the evening. There is ≥ 2 billion AFU per dose in total.
  Other Names: Akkermansia muciniphila (WB-STR-0001); Anaerobutyricum hallii (WB-STR-0008); Clostridium butyricum (WB-STR-006); Clostridium beijerinckii (WB-STR-0005); Bifidobacterium infantis (Dupont Danisco); chicory root inulin
  Arms: Probiotic
Other: Placebo — Ingredients include oligofructose, grape food color, magnesium stearate, silica and a delayed release capsule.
  Recommended storage is in a refrigerated environment at approximately 4°C. The product should not be frozen. It is recommended that the product be used within 2 months after opening the bottle. Participants are asked to take 2 capsules daily with food, 1 in the morning and 1 in the evening.
  Arms: Placebo

SUMMARY:
This study is a single center randomized control trial of a probiotic based intervention in pregnancies complicated by gestational diabetes. A healthy gut microbiome is now recognized as a key component of human health and dysbiosis of the gut microbiome, including lack of diversity, is believed to contribute to the development of many diseases and alter glucose control. The study aims to explore whether this probiotic intervention will improve glucose control and change the gut microbiome. Participants may be enrolled and randomized after diagnosis of gestational diabetes between 24 and 31 weeks gestation. 115 participants will be randomized in a ratio of 2 in the probiotic intervention group to 1 in the placebo group. Participants will stop taking the intervention at 6 weeks postpartum. At this time, they will be unblinded and offered the option of participating in an open-label extension of the intervention until 6 months postpartum.

DETAILED DESCRIPTION:
The chosen study design is a single-center, randomized, double-blind, parallel-group, placebo-controlled trial. Participants will be randomized by 2:1 to probiotic intervention or placebo. This is an exploratory study examining the impact of the intervention on glucose control among pregnant persons diagnosed with gestational diabetes.

Participants may be enrolled and randomized after diagnosis of GDM between 240 and 316 weeks gestation. Participants will stop taking the intervention at 6 weeks postpartum. At this time, they will be unblinded and offered the option of participating in an open-label extension of the intervention until 6 months postpartum.

Participants will be seen for up to 4 study visits: 3 mandatory visits in the main study and 1 in the optional extension. Brief visit outlines are below.

Visit 1 at 24-31 weeks gestation:

* eligibility confirmation
* consent
* randomization
* weight, height, blood pressure, method of glucose control from chart
* dispense investigational product
* baseline survey
* pregnancy history questionnaire
* Diet Screening for Adults in Canada (D-SAC)
* Automated Self-Administered 24-Hour Dietary Recall (ASA) x2
* Libre2 1 week of monitoring data
* concommitant medication log
* maternal rectal swab

Visit 2 at 37 weeks gestation:

* weight, height, blood pressure, method of glucose control from chart
* dispense and reconcile investigational product
* D-SAC
* ASA x2
* Libre2 1 week of monitoring data
* concommitant medication log
* maternal rectal swab
* adverse event log

Delivery:

* infant consent
* weight, height, blood pressure, method of glucose control from chart
* delivery chart review
* Libre2 1 week of monitoring data
* weigh placenta
* concommitant medication log
* adverse event log

Visit 3 at 6 weeks postpartum:

* reconcile investigational product
* unblind
* postpartum survey
* D-SAC
* ASA x2
* concommitant medication log
* maternal rectal swab
* infant fecal swab
* adverse event log
* study completion form

Optional Open Label Extension - At 6 weeks postpartum, once all study components are complete, participants will be unblinded and invited to participate in an open label, single arm extension of the intervention till 6 months postpartum. Participants who agree to participate in the extension of the intervention will be provided with additional open-label product until 6 months postpartum.

Visit E1 (open label extension, visit done with V3)

* enroll in extension if desired
* dispense open label product
* maternal and infant consent

Visit E2 at 6 months postpartum:

* Chart review
* D-SAC
* ASA x2
* concommitant medication log
* maternal rectal swab
* infant fecal swab
* adverse event log
* study completion form

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following inclusion criteria to be eligible for enrollment into the study:

1. Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
2. Participant has given written consent after study has been explained according to local regulatory requirements and before any study specific procedures.
3. Age ≥16 years at the time of consent.
4. Singleton pregnancy.
5. Live fetus (documented positive fetal heartbeat prior to recruitment)
6. Diagnosis of Gestational Diabetes (GDM) at the time of inclusion (documented 50g glucose challenge test (>11.1 mmol/L) and/or 75g oral glucose tolerance test with results exceeding the normal range (fasting >5.3 mmol/L, 1 hour >10.6 mmol/L, or 2 hour > 8.9 mmol/L)
7. Willing to provide fecal swab samples.
8. Willing to wear a continuous glucose monitor from enrollment until delivery and for 14 days at 6 weeks postpartum.
9. Willing to provide results from the continuous glucose monitor using the associated app on their mobile device.
10. Willing to complete surveys related to diet, pregnancy history, and health history.
11. Plan to reside in the study area at least until delivery and to deliver at Kingston Health Sciences Center (KHSC).
12. Willing to test for Group B Strep during pregnancy

Exclusion Criteria:

Any individual meeting any of the following criteria is not eligible for participation in this study:

1. Current diagnosis of severe gestational hypertension, preeclampsia, HELLP, intrauterine growth restriction, or other clinically significant pregnancy complication(s) at the time of enrollment.
2. Sustained use of substances, such as alcohol, cannabis, nicotine, and other recreational drugs. This is defined as any use after the patient is aware that they are pregnant OR as per the discretion of the investigator.
3. Systemic antibiotic or antifungal use ≤3 months prior to enrollment.
4. Active clinical infection(s), such as sexually transmitted infections, urinary tract infectionss, systemic infections, periodontal disease or positive blood cultures ≤3 months prior to enrollment
5. Acute or chronic clinically significant abnormality or poorly controlled pre-existent co-morbidities, such as autoimmune disease, inflammatory bowel disease (IBD), Crohn's, colitis, or other conditions, that, in the opinion of the investigator, might confound study results.
6. Prescription medications, especially relating to gastric function, or immunosuppressants, that, in the opinion of the investigator, might confound study results.
7. Known hypersensitivity to >4 first-line antimicrobial therapies against Akkermansia muciniphila, Clostridium beijerinckii, Clostridium butyricum, Anaerobutyricum hallii: Penicillin, Piperacillin, Tetracycline, Amoxicillin, Ampicillin.
8. Known hypersensitivity to >4 first-line antimicrobial therapies against Bifidobacterium infantis Bi-26TM: Gentamicin, Kanamycin, Streptomycin, Tetracycline, Erythromycin, Clindamycin, Ampicillin, Vancomycin.
9. Any conditions that, in the Investigator's judgement, may interfere with participant's ability to comply with study procedures or receipt of prenatal care, such as behavioural or cognitive impairment or neuropsychiatric illness.
10. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.
11. Pill swallowing phobia or inability to swallow pills.
12. Not taking any other probiotic supplements during the study intervention period.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control - Mean Fasting Glucose | 38th week of pregnancy (37+0-37+6 weeks gestation)
  To assess the impact that the probiotic based intervention has on glycemic control during pregnancy. Measured using continuous glucose monitoring comparing the week after randomization to the 38th week of pregnancy (37+0-37+6).
  Assessed based on:
  a) Mean fasting glucose over one week of continuous glucose monitoring.
Glycemic Control - Mean Glucose | 38th week of pregnancy (37+0-37+6 weeks gestation)
  To assess the impact that the probiotic based intervention has on glycemic control during pregnancy. Measured using continuous glucose monitoring comparing the week after randomization to the 38th week of pregnancy (37+0-37+6).
  Assessed based on:
  b) Mean glucose over one week of continuous glucose monitoring.
Glycemic Control - Time in Ranges | 38th week of pregnancy (37+0-37+6 weeks gestation)
  To assess the impact that the probiotic based intervention has on glycemic control during pregnancy. Measured using continuous glucose monitoring comparing the week after randomization to the 38th week of pregnancy (37+0-37+6).
  Assessed based on:
  c) Proportion of time in range (3.9-10.0 mmol/L), hypoglycemia (<3.9 mmol/L), severe hypoglycemia (<3.0 mmol/L), hyperglycemia (>10.0 mmol/L) and severe hyperglycemia (>13.9 mmol/L) over one week of continuous glucose monitoring.
Glycemic Control - HbA1C | 38th week of pregnancy (37+0-37+6 weeks gestation)
  To assess the impact that the probiotic based intervention has on glycemic control during pregnancy. Measured using continuous glucose monitoring comparing the week after randomization to the 38th week of pregnancy (37+0-37+6).
  Assessed based on:
  d) HbA1C

SECONDARY OUTCOMES:
Glycemic Therapy Requirements | At Delivery
  Explore whether therapy requirements such as insulin and/or metformin differ between the probiotic intervention and placebo groups.
Group B Strep | At Delivery
  Explore whether the prevalence of Group B Strep in late pregnancy differs between the probiotic intervention and placebo groups.
Pregnancy Outcomes - Gestational Age at Delivery | At Delivery
  Explore differences in gestational age at delivery.
Pregnancy Outcomes - Mode of Delivery | At Delivery
  Explore differences in mode of delivery.
Maternal Outcomes - Severe Maternal Morbidity | Within 42 days of delivery
  Explore differences in severe maternal morbidity within 42 days of delivery.
Maternal Outcomes - Weight Change | At Delivery
  Explore differences in maternal weight change.
Neonatal Outcomes - Birthweight | At delivery
  Explore differences in birthweight
Neonatal Outcomes - NICU Admissions | Within 28 days of delivery
  Explore differences in number of neontal intensive care unit admissions.
Neonatal Outcomes - Hypoglycemia | Within 72 hours of delivery.
  Explore differences in incidence of neonatal hypoglycaemia.
Maternal Gut Microbiome - Metagenome | 38th week of pregnancy, 6 weeks postpartum, 6 months postpartum
  To investigate if, and to what extent, the probiotic based intervention alters the gut metagenome. Sample will be collected via rectal swab for maternal participants.
Maternal Gut Microbiome - Metabolome | 38th week of pregnancy, 6 weeks postpartum, 6 months postpartum
  To investigate if, and to what extent, the probiotic based intervention alters the gut metabolome. Sample will be collected via rectal swab for maternal participants.
Infant Gut Microbiome - Metagenome | 6 Weeks of Age
  To investigate if, and to what extent, the probiotic based intervention alters the gut metagenome. For infant participants, swabs of stool samples will be used.
Infant Gut Microbiome - Metabolome | 6 Weeks of Age
  To investigate if, and to what extent, the probiotic based intervention alters the gut metabolome. For infant participants, swabs of stool samples will be used.
Safety & Side Effect Profile | Bi-weekly until 1 month after last dose is taken
  To document the safety, side effect profile of the probiotic and adherence to the intervention. Specific adverse events of interest include gastrointestinal discomfort, gas, or bloating, indigestion symptoms or mild stomach upset, diarrhea, constipation, and allergic reaction.

OTHER OUTCOMES:
Cardiometabolic Outcomes - HbA1C | 6 Months Postpartum
  Compare cardiometabolic outcomes at 6 months postpartum between based on probiotic exposure in pregnancy and/or postpartum, including HbA1C.
Cardiometabolic Outcomes - 2 Hour OGTT | 6 Months Postpartum
  Compare cardiometabolic outcomes at 6 months postpartum between based on probiotic exposure in pregnancy and/or postpartum, including 2-hour oral glucose tolerance test.
Cardiometabolic Outcomes - Lifetime CVR Score | 6 Months Postpartum
  Compare cardiometabolic outcomes at 6 months postpartum between based on probiotic exposure in pregnancy and/or postpartum, including lifetime cardiovascular risk score.
Cardiometabolic Outcomes - 30 Year CVR Score | 6 Months Postpartum
  Compare cardiometabolic outcomes at 6 months postpartum between based on probiotic exposure in pregnancy and/or postpartum, including 30 Year cardiovascular risk score.
Cardiometabolic Outcomes - Metabolic Syndrome | 6 Months Postpartum
  Compare cardiometabolic outcomes at 6 months postpartum between based on probiotic exposure in pregnancy and/or postpartum, including metabolic syndrome prevalence.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme N Smith, MD, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University & Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
After the 5 year data retention period the study database and data dictionary will be made available in a public data archive. This will likely be the Queen's University Library Research Data Archive in the Scholars Portal Dataverse. Further details will be provided as available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the 5 year data retention period the study database and data dictionary will be made available in a public data archive.
Access Criteria: Public data archive.